CLINICAL TRIAL: NCT01694056
Title: Soy Protein Intake and the Metabolic Syndrome: Reducing Inflammation to Improve Insulin Resistance and Glucose Homeostasis
Brief Title: Soy Protein Intake and the Metabolic Syndrome
Acronym: SOY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Alpro Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NL39991.081.12
Record Dates: First submitted 2012-09-04; First posted 2012-09-26 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soy protein diet (Experimental): High mixed protein diet (20 en%) with 25gr of soy protein per day
  Interventions: Other: Soy protein diet
- Control diet (Active Comparator): High mixed protein diet (20 en%)
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Soy protein diet — 4 weeks high protein diet (20 en%) with 25gr of soy protein per day
  Arms: Soy protein diet
Other: Control diet — 4 weeks high mixed protein diet (20 en%)
  Arms: Control diet

SUMMARY:
Soy protein has a high biological value, and contains several potential health-related nutritional factors, i.e. its amino acids pattern, biological active peptides and non-protein compounds such as isoflavones. In the field of obesity and blood lipids soy protein is well-studied and appreciated; it improves circulating blood lipids and is associated with weight reduction. The effect of soy on insulin resistance, glucose homeostasis and the metabolic syndrome is less frequently studied. However, several molecular mechanisms of action of soy protein make it a promising approach.

DETAILED DESCRIPTION:
Objective: The primary objective of the present study is to evaluate the effect of a high soy protein diet on insulin resistance and glycemic control in participants with characteristics of the metabolic syndrome. Secondly, the present study will evaluate whether reduced low-grade inflammation is a possible mechanism underlying the improvement in insulin resistance and glucose homeostasis. Finally, it will be assessed whether soy protein has beneficial effects on components of the metabolic syndrome, such as cardio-metabolic risk factors, blood lipid profile, blood pressure and endothelial function, fat storage in the liver and gene-expression in subcutaneous abdominal adipose tissue.

Study design: Single-blind, cross-over strictly-controlled dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 45-70 years
* No menstrual cycle for ≥1 year
* Stable body weight for ≥6 months (no weight gain/loss > 3 kg)
* Stable exercise habits during the last 6 months, and not participating in any vigorous exercise program
* Central obesity: waist circumference ≥80 cm

Plus any one of the following four factors:

* Raised triglyceride level: ≥1.7 mmol/L;
* Reduced high-density lipoprotein (HDL) cholesterol: <1.29 mmol/L
* Raised blood pressure: systolic blood pressure ≥135 mmHg or diastolic BP ≥85 mmHg or use of blood pressure lowering medication
* Raised fasting plasma glucose ≥ 5.6 mmol/L

Exclusion Criteria:

* (Undiagnosed) Diabetes - but not impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) as evaluated by an oral glucose tolerance test at screening
* Active hearth disease, i.e. history of myocardial infarction, stroke or angina pectoris
* Active or a history of thyroid disease
* Cancer or other malignancies in the past 5 years
* Two sided ovariectomy
* Drug use knowing to interfere with objectives of the study
* oral corticosteroids, lipid-lowering drugs (statins)
* anti-conceptive use (such as the pill or IUD)
* hormone replacement therapy
* long-term antibiotics use
* Habitual intake of soy foods (>1 soy food per week)
* Isoflavone supplements
* Vegetarian
* Following, or have recently followed a (weight-loss) diet
* Allergic to soy or dairy products
* Smoking
* Consuming more than 14 glasses of alcohol per week
* Donated or intended to donate blood 2 months before till two months after the study
* Participation in another biomedical study within 1 month before the first screening visit
* Not willing to be informed if deviations are found in blood samples
* Contraindications to MRI scanning

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 4 weeks
  Insulin sensitivity is measured with an intravenous glucose tolerance test (IVGTT).

SECONDARY OUTCOMES:
Adipose tissue gene expression | 4 weeks
  Adipose tissue samples will be collected for subsequent gene expression analysis.
Blood lipids | 4 weeks
  Circulating triglycerides, free fatty acids (FFA), and HDL and total cholesterol will be measured in fasted blood samples, LDL will be calculated.
Inflammation markers and adipokines | 4 weeks
  For low-grade inflammation interleukins, tumor necrosis factor-α, C-reactive protein and adipokines will be measured in fasting blood samples. Furthermore, peripheral blood mononuclear cells (PBMC's) will be collected to measure expression of genes involved in lipid handling and inflammation.
Cardio-metabolic risk factors | 4 weeks
  Blood pressure and macro vascular regional arterial stiffness will be assessed by Pulse Wave Analysis (PWA). Besides PWA, we will also measure markers for endothelial function in fasting blood samples.
Hepatic lipid content | 4 weeks
  Hepatic lipid content The lipid content in liver will be quantified by proton magnetic resonance spectroscopy (1H -MRS)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mensink, PhD, Study Chair — Departement of Human Nutrition, Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands

REFERENCES:
- [Derived] van Nielen M, Feskens EJ, Rietman A, Siebelink E, Mensink M. Partly replacing meat protein with soy protein alters insulin resistance and blood lipids in postmenopausal women with abdominal obesity. J Nutr. 2014 Sep;144(9):1423-9. doi: 10.3945/jn.114.193706. Epub 2014 Jul 9. PMID 25008579